CLINICAL TRIAL: NCT04268459
Title: Estimation of Benefit From Regular Versus Leakage-related Exchange of Voice Prosthesis in Patients Post Laryngectomy Considering Complications Rate, Fistula Colonization by Candida Species and Patients Satisfaction Feedback.
Brief Title: Estimation of Benefit From Regular Versus Leakage-related Exchange of Voice Prosthesis in Patients Post Laryngectomy.
Acronym: RvLPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Anna Rzepakowska, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1WF_CT_1_2020
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Laryngectomy; Voice; Prosthesis Failure
Keywords: voice prosthesis, laryngectomy, complications
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular exchange (Active Comparator): Patients will be appointed each 3 months for regular exchange of voice prosthesis.
  Interventions: Device: Provox prosthesis exchange
- Leakage exchange (Active Comparator): Patients will have voice prosthesis exchange when leakage occurs.
  Interventions: Device: Provox prosthesis exchange

INTERVENTIONS:
Device: Provox prosthesis exchange — Each patient post laryngectomy will be randomly assigned to one arm of intervention. The voice prosthesis exchange in all patients will be performed in local anaesthesia. The microbiological samples with cotton swabs will be collected from tracheoesophageal fistula on prosthesis exchange. The clinical evaluation and patients satisfaction from prosthesis usage will be performed on each exchange.

SUMMARY:
The tracheoesophageal voice with voice prosthesis is currently the mainstay of voice rehabilitation post laryngectomy. The primary surgical technique of tracheoesophageal fistula formation with insertion of prosthesis and quick and easy process of voice rehabilitation are main encouraging factors. However, the usage of the prosthesis relates to a significant number of complications rated from 10 to 60%. The most common reported complication is transprosthetic leakage that determines the need of device exchange. However in some patients occur more serious complications eg. periprosthetic leakage, granulation or atrophy of mucosa around the fistula, dislocation of prosthesis, that may require anti-inflammatory treatment, temporary nasogastric tube feeding or surgical procedure. The standard protocol is voice prosthesis exchange due to transprosthetic leakage. Optionally the device could be replaced regularly to prevent both transprosthetic leakage and other complication occurrence.

In the study we plan to compare the benefits from regular (each three month) versus leakage-related exchange of voice prosthesis post laryngectomy including the rate of complications, fistula colonization by Candida species and patients feedback.

ELIGIBILITY:
Inclusion Criteria:

* patients post laryngectomy with primary insertion of voice prosthesis

Exclusion Criteria:

* patients post laryngopharyngectomy with digestive tract reconstruction with jejunum of free flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-10 (Estimated); Primary Completion 2021-03-10 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of complications rate. | Control will be continued for 12 months post laryngectomy.
  In both arms of the study we will compare the incidence of following complications: periprosthetic leakage, granulation or atrophy of mucosa around the fistula, dislocation of prosthesis

SECONDARY OUTCOMES:
Fistula colonization with Candida species. | Control will be continued for 12 months post laryngectomy.
  We will compare microbiological results on subsequent prosthesis exchanges in both arms.
Prosthesis replacement scheme and patient satisfaction. | Control will be continued for 12 months post laryngectomy.
  On each voice prosthesis exchange patients will be asked three questions, assessed with Visual Analog Scale, on their feedback on voice prosthesis use, procedure of prosthesis replacement and voice quality.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rzepakowska, PhD, Study Chair — Medical University of Warsaw
Locations (1):
- Department of Otorhinolaryngology, Head andNeck Surgery of Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Date will become available from April 2022 until April 2023.
Access Criteria: on request

REFERENCES:
- [Derived] Zurek M, Czesak M, Majszyk D, Rzepakowska A. Benefit from regular versus leakage-related exchange of voice prostheses in patients post-laryngectomy considering complication rates and patient satisfaction feedback-a randomized case-controlled trial. Front Oncol. 2025 Jan 24;15:1468955. doi: 10.3389/fonc.2025.1468955. eCollection 2025. PMID 39926276
- [Derived] Zurek M, Czesak M, Czerwinska ME, Berezovska D, Niemczyk K, Rzepakowska A. A double-blind randomized clinical trial of inflammatory cytokine and pepsin levels in the saliva of patients with voice prostheses. Head Neck. 2024 Sep;46(9):2116-2122. doi: 10.1002/hed.27847. Epub 2024 Jun 12. PMID 38864228